CLINICAL TRIAL: NCT03743246
Title: A Phase 1/2, Open-label, Single Arm, Multicohort, Multicenter Trial to Evaluate the Safety and Efficacy of JCAR017 in Pediatric Subjects With Relapsed/Refractory (r/r) B-cell Acute Lymphoblastic Leukemia (B-ALL) and B-cell Non-Hodgkin Lymphoma (B-NHL).
Brief Title: A Study to Evaluate the Safety and Efficacy of JCAR017 in Pediatric Subjects With Relapsed/Refractory (r/r) B-cell Acute Lymphoblastic Leukemia (B-ALL) and B-cell Non-Hodgkin Lymphoma (B-NHL)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Absence of significant therapeutic benefit over existing therapies
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCAR017-BCM-004; U1111-1220-3324 (Registry Identifier: WHO); 2018-001246-34 (EudraCT Number)
Record Dates: First submitted 2018-10-18; First posted 2018-11-16 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin
Keywords: Pediatric; JCAR017; CAR-T; CART; CD19; ALL; NHL; DLBCL; BL; PMBCL; Cell Therapy; LisoCell; Young Adults; Lymphoproliferative disorders; Immune system diseases; Leukemia; Lymphoma; lymphatic diseases
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Immune System Diseases; Leukemia; Lymphoma; Lymphatic Diseases | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of JCAR017 (Experimental): Subjects will receive Lymphodepleting chemotherapy with intravenous (IV) fludarabine (30 mg/m2/day for 3 days) plus cyclophosphamide IV (300 mg/m2/day for 3 days) (flu/cy) concurrently, followed by JCAR017 cells infusion. Phase 1 will evaluate up to 5 JCAR017 cells dose levels and dose escalation/de-escalation will follow a modified toxicity probability interval (mTPI-2) algorithm. The declared RP2D in Phase 1 will be applied to the subjects enrolled in Phase 2
  Interventions: Drug: JCAR017; Drug: Lymphodepleting; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: JCAR017 — JCAR017
Drug: Lymphodepleting — Lymphodepleting
Drug: Fludarabine — Fludarabine
Drug: Cyclophosphamide — Cyclophosphamide

SUMMARY:
This is a Phase 1/2, open-label, single arm, multicohort study to evaluate the safety and efficacy of JCAR017 in pediatric subjects aged ≤ 25 years with CD19+ r/r B-ALL and B-NHL.

Phase 1 will identify a recommended Phase 2 dose (RP2D). Phase 2 will evaluate the efficacy of JCAR017 RP2D in the following three disease cohorts: Cohort 1 (r/r B-ALL), Cohort 2 (MRD+ B-ALL) and Cohort 3 (r/r B-NHL, [DLBCL, BL, or PMBCL]). A Simon's Optimal two-stage study design will be applied to Cohort 1 and 2 in Phase 2.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, single arm, multicohort study incorporating Simon's Optimal two-stage design to evaluate the safety and efficacy of JCAR017 in pediatric subjects aged ≤ 25 years with CD19+ r/r B-ALL and B-NHL.

In the Phase 1, up to 5 dose levels will be of JCAR017 will be evaluated. Enrollment will commence in pediatric subjects with r/r B-ALL at Dose Level 1 (DL1) of 0.05x10^6 CAR+ T cells/kg (maximum DL1 of 5x10^6 JCAR017 CAR+ T cells [non-weight adjusted]). If this dose is confirmed to be safe and tolerable, additional subjects will be enrolled at higher dose(s) up to 0.75 x10^6 CAR+ T cells/kg (maximum of 75x10^6 JCAR017 CAR+ T cells [non-weight adjusted]) with the aim to identify the RP2D. Dose escalation/de-escalation will follow a modified toxicity probability interval (mTPI-2) algorithm. A Safety Review Committee (SRC) will recommend the Phase 2 dose (defined as RP2D) based on an integrated assessment of the safety, PK and preliminary efficacy information from at least 10 pediatric subjects treated at the RP2D.

In Phase 2, a minimum of 71 additional subjects (< 18 years of age) will be enrolled into one of the 3 cohorts listed below. The sample size for Cohorts 1 and 2 is calculated according to Simon's Optimal two-stage design. The 10 or more pediatric subjects treated at the RP2D in Phase 1 will form part of the sample size (ie, Cohort 1 and Cohort 2). Therefore, the protocol intends to treat 81 primary endpoint evaluable pediatric subjects in Phase 2, if warranted by the evaluation of results at the completion of the first stage of the study in each cohort.

* Cohort 1 (r/r B-ALL): 48 evaluable pediatric subjects (13 subjects in Stage 1 and 35 in Stage 2)
* Cohort 2 (MRD+ B-ALL): 23 evaluable pediatric subjects (9 subjects in Stage 1 and 14 subjects in Stage 2)
* Cohort 3 (r/r B-NHL [DLBCL, BL, or PMBCL]): 10 evaluable pediatric subjects. Due to the very low incidence rate and therefore expected low subject accrual, there is no formal sample size for this arm.

Up to 20 additional B-ALL subjects between 18 and 25 years of age may be enrolled in Phase 2.

Following treatment with JCAR017 subjects will then enter the post-treatment period for disease progression/relapse, safety, CAR T cell persistence, and survival up to 24 months after administration of JCAR017.

Efficacy will be assessed both locally and by an Independent Review Committee. Response assessments will be based on bone marrow and blood morphologic criteria, physical examination findings, along with laboratory assessments of cerebral spinal fluid (CSF) and bone marrow MRD (B-ALL only) assessments. B-NHL subjects will also have radiographic disease assessment by CT/MRI scans and tumor biopsies, if accessible.

Post-study follow-up for survival, relapse, long-term toxicity, and lentiviral vector safety will continue under a separate long-term follow-up protocol for up to 15 years after the JCAR017 infusion as per health authority regulatory guidelines.

An Independent Data Monitoring Committee will monitor the study conduct.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Phase 1: Subject < 18 years of age and weighs ≥ 6 kg at the time of signing the informed consent form (ICF)/informed assent form (IAF).

   Phase 2: Subject ≤ 25 years of age and weighs ≥ 6 kg at the time of signing the ICF/IAF.
2. Subject (when applicable, parental/legal representative) must understand and voluntarily provide permission to the ICF/IAF prior to conducting any study-related assessments/procedures.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Investigator considers the subject is appropriate for adoptive T cell therapy.
5. Evidence of CD19 expression via flow cytometry (peripheral blood or bone marrow) or immunohistochemistry (bone marrow biopsy)
6. Subject has a Karnofsky score of ≥ 50 (subjects ≥ 16 years of age) or a Lansky score ≥ 50 (subjects < 16 years of age).
7. Diagnosis of B-cell ALL or B-cell NHL as defined below:

   Phase 1: Subjects with r/r B-ALL, defined as morphological evidence of disease in BM (5% or greater lymphoblast by morphology) and either of the following:
   * First or greater marrow relapse, or
   * Any marrow relapse after allogeneic HSCT, or
   * Primary refractory defined as not achieving a CR or a CRi after 2 or more separate induction regimens (or chemo-refractory as not achieving CR/CRi after 1 cycle of standard chemotherapy for relapsed leukemia), or
   * Ineligible for allogeneic HSCT Note: Subjects will be included regardless of MRD status.

   Phase 2: Subjects with one of the following:
   * Cohort 1: r/r B-ALL, defined as morphological evidence of disease in BM (5% or greater lymphoblast by morphology) and either:

     * First or greater marrow relapse, or
     * Any marrow relapse after allogeneic HSCT, or
     * Primary refractory defined as not achieving a CR or a CRi after 2 or more separate induction regimens (or chemo-refractory as not achieving CR/CRi after 1 cycle of standard chemotherapy for relapsed leukemia), or
     * Ineligible for allogeneic HSCT.
   * Cohort 2: MRD+ B-ALL, defined as:

     * < 5% lymphoblasts by morphology with,
     * MRD detected by a validated assay at a frequency of 1 x10-4 or greater in BM cells. Subjects eligible for enrollment in Cohort 2 are those with MRD positive morphologic CR2 after re-induction when these subjects had previously experienced an early relapse (< 36 months) after first-line chemotherapy. Subjects who are in MRD+ morphologic CR3 and later, regardless of time to relapse in earlier lines, are also eligible. Subjects who are in morphologic relapse at screening (r/r B-ALL) and become MRD+ after bridging chemotherapy are also eligible for treatment in Cohort 2.
   * Cohort 3: r/r B-NHL (DLBCL, BL or PMBCL), defined as measurable disease after 1 or more lines of chemotherapy and/or having failed HSCT or being ineligible for HSCT.

   Note: B-NHL subjects with secondary CNS lymphoma involvement are eligible however subject selection must consider clinical risk factors for severe neurological AEs and alternative treatment options. Subjects should only be enrolled if the Investigator considers the potential benefit outweighs the risk for the subject.
8. Subjects with Philadelphia chromosome positive ALL are eligible if they are intolerant to or have failed one or more lines of tyrosine-kinase inhibitor (TKI) therapy or if TKI therapy is contraindicated.
9. Adequate organ function, defined as:

   * Adequate BM function to receive LD chemotherapy as assessed by the Investigator.
   * Subject with adequate renal function, which is defined as:

   Serum creatinine based on age/gender as described below. Subjects that do not meet the criteria but who have a creatinine clearance or radioisotope glomerular filtration rate (GFR) > 70 mL/min/1.73 m2 are eligible.• Alanine aminotransferase (ALT) ≤ 5 x upper limit of normal (ULN) and total bilirubin < 2.0 mg/dL (or < 3.0 mg/dL for subjects with Gilbert's syndrome or leukemic/lymphomatous infiltration of the liver).
   * Adequate pulmonary function, defined as ≤ Grade 1 dyspnea according to Common Toxicity Criteria for Adverse Events (CTCAE) and oxygen saturation (SaO2) ≥ 92% on room air.
   * Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) ≥ 40% as assessed by echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) within 4 weeks prior to leukapheresis.
10. Adequate vascular access for leukapheresis procedure.
11. Participants must agree to use effective contraception

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject with a history of another primary malignancy that has not been in remission for at least 2 years prior to enrollment.
5. Subjects who have received previous CD19-targeted therapy must have CD19-positive disease confirmed since completing the prior CD19-targeted therapy.
6. Prior CAR T cell or other genetically-modified T cell therapy.
7. Subject with a previous history of or active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection.
8. Subjects with uncontrolled systemic fungal, bacterial, viral or other infection (including tuberculosis) despite appropriate antibiotics or other treatment at the time of leukapheresis or JCAR017 infusion.
9. Subject has presence of acute or chronic graft-versus-host disease (GVHD).
10. Subject with active autoimmune disease requiring immunosuppressive therapy.
11. Subject has cardiac disorders (CTCAE version 4.03 Grade 3 or 4) within the past 6 months.
12. Subject with a concomitant genetic syndrome, with the exception of Down's syndrome.
13. Subject with active CNS disease and significant neurological deterioration. Subjects with CNS-2 or CNS-3 involvement are eligible provided they are asymptomatic and do not have significant neurological deterioration and, in the opinion of the study investigator, the CNS disease burden can be controlled until JCAR017 infusion.
14. Subject with a history or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, cerebral edema, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
15. Subject is pregnant or nursing.
16. Subject has used the following:

    * Therapeutic doses of corticosteroids (defined as > 0.4 mg/kg maximum 20 mg/day prednisone or equivalent) within 7 days prior to leukapheresis or 72 hours prior to JCAR017 infusion. Physiologic replacement, topical, and inhaled steroids are permitted.
    * Low-dose chemotherapy (eg, vincristine, rituximab, cyclophosphamide ≤ 300 mg/m2) given after leukapheresis to maintain disease control must be stopped ≥ 7 days prior to LD chemotherapy.
    * Cytotoxic chemotherapeutic agents that are not considered lymphotoxic within 1 week prior to leukapheresis. Oral anticancer agents are allowed if at least 3 half-lives have elapsed prior to leukapheresis.
    * Lymphotoxic chemotherapeutic agents (eg, cyclophosphamide, ifosfamide, bendamustine) within 2 weeks prior to leukapheresis.
    * Experimental agents within 4 weeks prior to leukapheresis unless no response or PD is documented on the experimental therapy and at least 3 half-lives have elapsed prior to leukapheresis.
    * Immunosuppressive therapies within 4 weeks prior to leukapheresis and JCAR017 infusion (eg, calcineurin inhibitors, methotrexate or other chemotherapeutics, mycophenolate, rapamycin, thalidomide, immunosuppressive antibodies such as antitumor necrosis factor [TNF], anti-IL-6, or anti-IL-6R).
    * Donor lymphocyte infusions (DLI) within 6 weeks prior to JCAR017 infusion.
    * Radiation within 6 weeks prior to leukapheresis. Subjects must have PD in irradiated lesions or have additional non-irradiated lesions to be eligible. Radiation to a single lesion, if additional non-irradiated, measurable lesions are present, is allowed up to 2 weeks prior to leukapheresis.
    * Allogeneic HSCT within 90 days prior to leukapheresis.
17. Tumor invasion of venous or arterial vessels (B-NHL subjects only).
18. Deep Venous Thrombosis (DVT) or Pulmonary Embolism (PE) within 3 months prior to leukapheresis. Subjects with DVT or PE that occurred longer than 3 months prior to leukapheresis, who still require ongoing therapeutic levels of anti-coagulation therapy, are also excluded.
19. Existence of CD19-negative clone(s) of leukemia cells

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (9):
  - Local Institution - 163, Duarte, California
  - Local Institution - 167, Redwood City, California
  - Local Institution - 166, St. Petersburg, Florida
  - Local Institution - 160, New York, New York
  - Local Institution - 162, Philadelphia, Pennsylvania
  - Local Institution - 164, Dallas, Texas
  - Local Institution - 165, Houston, Texas
  - Local Institution - 161, Seattle, Washington
  - Local Institution - 168, Wauwatosa, Wisconsin
- France (3):
  - Local Institution - 601, Lyon
  - Local Institution - 602, Marseille
  - Local Institution - 600, Paris
- Germany (2):
  - Local Institution - 501, Berlin
  - Local Institution - 500, Frankfurt
- Italy (2):
  - Local Institution - 301, Monza
  - Local Institution - 300, Roma
- Local Institution - 400, Utrecht, Netherlands
- Spain (2):
  - Local Institution - 251, Esplugues de Llobregat
  - Local Institution - 250, Madrid

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT03743246.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated and hence participants were not enrolled in Phase 2 cohorts (r/r B-ALL; MRD+ B-ALL; r/r B-NHL).
Groups:
- 0.05 x 10^6 CAR+ T Cells/kg: Participants with CD19+ relapsed/refractory (r/r) B-cell acute lymphoblastic leukemia (B-ALL) were infused with 0.05 x 10^6 CAR+ T cells per kilogram (kg) post leukapheresis.
- 0.15 x 10^6 CAR+ T Cells/kg: Participants with CD19+ relapsed/refractory (r/r) B-cell acute lymphoblastic leukemia (B-ALL) were infused with 0.15 x 106 CAR+ T cells/kg post leukapheresis.
- 0.50 x 106 CAR+T Cells/kg: Participants with CD19+ relapsed/refractory (r/r) B-cell acute lymphoblastic leukemia (B-ALL) were infused with 0.50 x 106 CAR+T cells/kg post leukapheresis.
- Not Assigned: Participants only underwent leukapheresis.
Period: Pre-Treatment Period
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg | Not Assigned
Started (Leukapheresed) | 9 | 8 | 3 | 1
Completed | 8 | 7 | 1 | 0
Not Completed | 1 | 1 | 2 | 1
Not completed — Failure to meet treatment criteria | 0 | 0 | 2 | 0
Not completed — Death | 0 | 1 | 0 | 1
Not completed — Study Drug Manufacturing Failure | 1 | 0 | 0 | 0
Period: Lymphodepleting Chemotherapy
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg | Not Assigned
Started | 8 | 7 | 1 | 0
Completed | 7 | 7 | 1 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0 | 0
Period: Treatment Period (JCAR017 Infusion)
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg | Not Assigned
Started | 7 (7 participant received conforming JCAR017 Infusion) | 7 (1 participant received non-conforming JCAR017 Infusion and 6 received conforming JCAR017 Infusion) | 1 (1 participant received conforming JCAR017 Infusion) | 0
Completed | 3 | 6 | 1 | 0
Not Completed | 4 | 1 | 0 | 0
Not completed — Other Reason | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg | Not Assigned | Total
Number analyzed (Participants) | 9 | 8 | 3 | 1 | 21
Age, Customized [Number; unit: participants]
  < 6 years | 3 | 4 | 2 | 0 | 9
  >= 6 to < 12 years | 5 | 3 | 1 | 0 | 9
  >= 12 to < 18 years | 1 | 1 | 0 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 2 | 0 | 11
  Male | 4 | 4 | 1 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 1 | 1 | 9
  Not Hispanic or Latino | 4 | 4 | 2 | 0 | 10
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 5 | 3 | 0 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events up to 30 Days Post JCAR017 Infusion
Description: An AE is defined as any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. Treatment Emergent Adverse Events (TEAEs) are defined as any AE occurring or worsening on the day of the JCAR017 infusion until 30 days post-treatment (JCAR017 infusion) using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 or greater.
Time Frame: From first JCAR017 infusion (Day 1) to 30 days after JCAR017 infusion
Population: Safety Analysis Set included all participants who received conforming JCAR017 infusion with baseline and post-baseline measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 7 | 6 | 1
Participants | 7 | 6 | 1

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: A DLT was defined as:
  * Death not related to disease progression
  * Grade (Gr) 4 (Life-threatening) neurotoxicity
  * Gr 3 (Severe) neurotoxicity of greater than 7 days
  * Gr 3 neurotoxicity does not revert to baseline within 28 days of the start date of the Grade 3 event
  * Seizures of grade that do not resolve within 7 days
  * Gr 4 cytokine release syndrome (CRS) that does not resolve to Grade ≤ 3 within 3 days
  * Gr 3 CRS that does not resolve to Grade ≤ 2 within 7 days
  * Any increase in aspartate aminotransferase (AST) or ALT > 3 × ULN and concurrent increase in total bilirubin > 2 × ULN that is unrelated to CRS and has no other probable reason to explain the combination of increases
  * Any cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic Gr 3 or 4 event not pre-existing or not due to the underlying malignancy
  * Any other Gr 3 or 4 event deemed unexpected by the Investigator and considered a DLT upon evaluation by the safety review committee
Time Frame: From first JCAR017 infusion (Day 1) to 28 days after JCAR017 infusion
Population: Dose-Limiting Toxicity Analysis Set included all participants who received conforming JCAR017 infusion and completed 28 days post JCAR017 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 5 | 5 | 1
Participants | 0 | 2 | 1

3. Primary Outcome: Concentration of JCAR017 in Peripheral Blood at Day 28 Post JCAR017 Infusion
Description: Concentration of JCAR017 in Peripheral Blood was assessed by droplet digital polymerase chain reaction.
Time Frame: At day 28 post JCAR017 infusion
Population: The PK Analysis Set include all participants who received JCAR017 infusion and have at least one measurable JCAR017 concentration. Participants available at specific timepoints have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies per microgram
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 3 | 3 | 1
copies per microgram | 1131.821 (64.658) | 1457.591 (75.558) | 2847.910 (NA) — Geometric coefficient of variation is not applicable as only a single participant was analyzed.

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events up to 90 Days Post JCAR017 Infusion
Description: An AE is defined as any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. Treatment Emergent Adverse Events (TEAEs) are defined as any AE occurring or worsening on the day of the JCAR017 infusion until 90 days post-treatment (JCAR017 infusion) using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 or greater. The following scale for grading was used - Grade 3 = Severe, Grade 4 = Life-Threatening.
Time Frame: From first JCAR017 infusion (Day 1) to 90 days after JCAR017 infusion
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 7 | 6 | 1
Participants
  At least one TEAE | 7 | 6 | 1
  At least one grade 3/4 TEAE | 6 | 5 | 1
  At Least One TEAE Related To JCAR017 | 5 | 5 | 1
  At Least One grade 3/4 TEAE Related To JCAR017 | 3 | 4 | 1

5. Secondary Outcome: Number of Participants With Serious Treatment-Emergent Adverse Events up to 90 Days Post JCAR017 Infusion
Description: Serious adverse events (SAE) are defined as any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/ birth defect; constitutes an important medical event. Treatment Emergent Adverse Events (TEAEs) are defined as any AE occurring or worsening on the day of the JCAR017 infusion until 90 days post-treatment (JCAR017 infusion) using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 or greater.
Time Frame: From first JCAR017 infusion (Day 1) to 90 days after JCAR017 infusion
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 7 | 6 | 1
Participants
  AT Least one Serious TEAE | 5 | 3 | 1
  At Least One Serious TEAE Related To JCAR017 | 1 | 3 | 1

6. Secondary Outcome: Change From Baseline at Day 28 in Hematology Laboratory Parameters- Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: Baseline is defined as the last assessment with non-missing value on or prior to the first date of the lymphodepletion chemotherapy.
Time Frame: Baseline and at Day 28
Population: Safety Analysis Set included all participants who received conforming JCAR017 infusion with baseline and post-baseline measurements. Participants available at specific timepoints have been analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 5 | 1
10^9 cells/L
  Basophils | 0.00 (0.025) | -0.01 (0.023) | -0.01 (NA) — Not applicable as only a single participant was analyzed.
  Eosinophils | 0.03 (0.048) | 0.08 (0.114) | -0.08 (NA) — Not applicable as only a single participant was analyzed.
  Leukocytes | 4.01 (8.338) | 0.59 (1.753) | -2.00 (NA) — Not applicable as only a single participant was analyzed.
  Lymphocytes | -0.22 (0.879) | 0.27 (1.286) | -0.57 (NA) — Not applicable as only a single participant was analyzed.
  Monocytes | 0.11 (0.163) | 0.09 (0.173) | -0.22 (NA) — Not applicable as only a single participant was analyzed.
  Neutrophils: number analyzed (Participants) | 5 | 4 | 1
  Neutrophils | 0.41 (0.782) | -0.18 (0.735) | -1.50 (NA) — Not applicable as only a single participant was analyzed.
  Platelets | 27.33 (132.672) | -68.60 (168.583) | -163.00 (NA) — Not applicable as only a single participant was analyzed.

7. Secondary Outcome: Change From Baseline at Day 28 in Hematology Laboratory Parameters- Basophils/Leukocytes; Eosinophils/Leukocytes; Lymphocytes/Leukocytes; Neutrophils/Leukocytes; Monocytes/Leukocytes
Description: as for outcome 6
Time Frame: Baseline and at Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 5 | 1
Ratio
  Basophils/Leukocytes | 0.25 (0.885) | -0.24 (0.654) | -0.30 (NA) — Not applicable as only a single participant was analyzed.
  Eosinophils/Leukocytes | 0.85 (1.402) | 4.28 (5.389) | -2.90 (NA) — Not applicable as only a single participant was analyzed.
  Lymphocytes/Leukocytes | -29.57 (21.690) | -16.30 (25.140) | 33.80 (NA) — Not applicable as only a single participant was analyzed.
  Neutrophils/Leukocytes | 26.45 (26.815) | 10.70 (18.797) | -33.90 (NA) — Not applicable as only a single participant was analyzed.
  Monocytes/Leukocytes | 4.35 (10.123) | 1.74 (4.515) | 0.20 (NA) — Not applicable as only a single participant was analyzed.

8. Secondary Outcome: Change From Baseline at Day 28 in Hematology Laboratory Parameters- Erythrocytes
Description: as for outcome 6
Time Frame: Baseline and at Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 5 | 1
10^12 cells/L | 0.04 (0.781) | 0.08 (0.268) | -0.70 (NA) — Not applicable as only a single participant was analyzed.

9. Secondary Outcome: Change From Baseline at Day 28 in Hematology Laboratory Parameters- Hematocrit
Description: as for outcome 6
Time Frame: Baseline and at Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: proportion of red blood cells in blood
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 5 | 1
proportion of red blood cells in blood | 0.00 (0.068) | 0.02 (0.016) | -0.03 (NA) — Not applicable as only a single participant was analyzed.

10. Secondary Outcome: Change From Baseline at Day 28 in Hematology Laboratory Parameters- Hemoglobin
Description: as for outcome 6
Time Frame: Baseline and at Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 5 | 1
grams per liter | 2.33 (24.312) | 6.20 (6.834) | -13.00 (NA) — Not applicable as only a single participant was analyzed.

11. Secondary Outcome: Change From Baseline at Day 28 in Chemistry Laboratory Parameters- Alanine Aminotransferase; Alkaline Phosphatase; Aspartate Aminotransferase; Lactate Dehydrogenase
Description: as for outcome 6
Time Frame: Baseline and at Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 5 | 1
units per liter
  Alanine aminotransferase | 5.33 (19.439) | 4.50 (16.299) | -19.00 (NA) — Not applicable as only a single participant was analyzed.
  Alkaline phosphatase: number analyzed (Participants) | 6 | 4 | 1
  Alkaline phosphatase | 53.50 (158.322) | 78.75 (40.950) | -121.00 (NA) — Not applicable as only a single participant was analyzed.
  Aspartate aminotransferase: number analyzed (Participants) | 6 | 4 | 1
  Aspartate aminotransferase | 29.17 (72.204) | 11.50 (13.675) | -1.00 (NA) — Not applicable as only a single participant was analyzed.
  Lactate dehydrogenase: number analyzed (Participants) | 6 | 4 | 1
  Lactate dehydrogenase | 992.33 (2238.888) | 22.25 (43.684) | -36.00 (NA) — Not applicable as only a single participant was analyzed.

12. Secondary Outcome: Change From Baseline at Day 28 in Laboratory Parameters- Albumin; Protein
Description: as for outcome 6
Time Frame: Baseline and at Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 4 | 1
grams per liter
  Albumin | 5.83 (9.663) | 6.75 (2.062) | -3.00 (NA) — Not applicable as only a single participant was analyzed.
  Protein | 4.00 (12.602) | 5.00 (6.683) | -6.00 (NA) — Not applicable as only a single participant was analyzed.

13. Secondary Outcome: Change From Baseline at Day 28 in Chemistry Laboratory Parameters- Bicarbonate; Blood Urea Nitrogen; Calcium; Chloride; Glucose; Magnesium; Phosphate; Potassium; Sodium, Triglyceride
Description: as for outcome 6
Time Frame: Baseline and at Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 4 | 1
mmol/L
  Bicarbonate | 2.53 (4.453) | -2.65 (1.919) | 4.10 (NA) — Not applicable as only a single participant was analyzed.
  Blood Urea Nitrogen | 3.60 (3.542) | 2.43 (0.826) | 0.20 (NA) — Not applicable as only a single participant was analyzed.
  Calcium | 0.13 (0.157) | 0.04 (0.058) | -0.17 (NA) — Not applicable as only a single participant was analyzed.
  Chloride | -1.50 (4.324) | 1.50 (1.291) | 1.00 (NA) — Not applicable as only a single participant was analyzed.
  Glucose | 0.32 (0.641) | -0.08 (0.472) | 14.90 (NA) — Not applicable as only a single participant was analyzed.
  Magnesium | 0.06 (0.107) | 0.06 (0.109) | 0.00 (NA) — Not applicable as only a single participant was analyzed.
  Phosphate | 0.02 (0.281) | -0.02 (0.336) | -0.16 (NA) — Not applicable as only a single participant was analyzed.
  Potassium | -0.05 (0.672) | 0.20 (0.535) | 1.50 (NA) — Not applicable as only a single participant was analyzed.
  Sodium | 1.00 (2.608) | 2.25 (2.217) | 2.00 (NA) — Not applicable as only a single participant was analyzed.
  Triglyceride | 0.45 (1.652) | 0.29 (0.320) | 0.33 (NA) — Not applicable as only a single participant was analyzed.

14. Secondary Outcome: Change From Baseline at Day 28 in Chemistry Laboratory Parameters- Bilirubin; Creatinine; Direct Bilirubin; Urate
Description: as for outcome 6
Time Frame: Baseline and at Day 28
Population: as for outcome 6
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 5 | 1
umol/L
  Bilirubin: number analyzed (Participants) | 6 | 4 | 1
  Bilirubin | 20.26 (41.498) | -1.00 (6.928) | 2.00 (NA) — Not applicable as only a single participant was analyzed.
  Creatinine: number analyzed (Participants) | 6 | 4 | 1
  Creatinine | 9.84 (14.218) | 1.50 (9.000) | -2.00 (NA) — Not applicable as only a single participant was analyzed.
  Direct Bilirubin: number analyzed (Participants) | 6 | 4 | 1
  Direct Bilirubin | 13.44 (33.601) | -0.25 (0.500) | 0.00 (NA) — Not applicable as only a single participant was analyzed.
  Urate: number analyzed (Participants) | 6 | 4 | 1
  Urate | 43.51 (94.081) | 85.00 (71.615) | 9.00 (NA) — Not applicable as only a single participant was analyzed.

15. Secondary Outcome: Number of Participants With Manufacturing Success of JCAR017 Product
Description: Successful product was defined as JCAR017 product was generated and able to be QC released (including nonconforming product) for infusion. Unsuccessful product is defined as no JCAR017 product could be generated after two manufacturing attempts using a single apheresis product for starting material or product was unable to be QC released for infusion.
Time Frame: From screening to JCAR017 infusion (day -35 to day 1)
Population: Pre-Treatment Set included all participants who have screened successfully into the study and underwent leukapheresis.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg | Not Assigned
Number analyzed (Participants) | 9 | 8 | 3 | 1
Participants | 7 | 7 | 2 | 1

16. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved either a complete response (CR) or complete response with incomplete blood recovery (CRi) on Day 28 that is confirmed on Day 56. Response assessment was performed according to the 2019 Comprehensive Cancer Network (NCCN) response criteria guidelines for pediatric acute lymphoblastic leukemia (ALL). CR is defined as absence of circulating blasts, extramedullary disease, lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement, Trilineage hematopoiesis (TLH) and < 5%, Absolute neutrophil count (ANC) > 1000 per microliter, Platelets > 100,000 per microliter and no recurrence for 4 weeks. CRi is defined as meeting all criteria for CR except platelets < 100,000/μL or ANC is < 1000/μL.
Time Frame: Up to Day 56
Population: Efficacy Analysis Set included all participants who fulfilled all study eligibility criteria, received conforming JCAR017 infusion, who did not demonstrate morphological remission at screening and who are not MRD negative upon restaging prior to initiation of lymphodepleting (LD) chemotherapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 4 | 1
percentage of participants | 50.0 [11.8 to 88.2] | 25.0 [0.6 to 80.6] | 100.0 [2.5 to 100.0]

17. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as time from first response (either CR or CRi) until progressive disease (PD), disease relapse, or death from any cause, whichever occurs first. Response assessment was performed according to the 2019 Comprehensive Cancer Network (NCCN) response criteria guidelines for pediatric ALL. CR is defined as absence of circulating blasts, extramedullary disease, lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement, Trilineage hematopoiesis (TLH) and < 5%, Absolute neutrophil count (ANC) > 1000 per microliter, Platelets > 100,000 per microliter and no recurrence for 4 weeks. CRi is defined as meeting all criteria for CR except platelets < 100,000/μL or ANC is < 1000/μL. Disease progression is defined as increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease.
Time Frame: From first response (either CR or CRi) until progressive disease (PD), disease relapse, or death from any cause, whichever occurs first (Up to approximately 14 months)
Population: Efficacy Analysis Set included all participants who fulfilled all study eligibility criteria, received conforming JCAR017 infusion, who did not demonstrate morphological remission at screening and who are not MRD negative upon restaging prior to initiation of lymphodepleting (LD) chemotherapy. Responders (either CR or CRi) are included in the analysis. Censored participants were also analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 3 | 1 | 1
months | 13.70 [2.46 to 13.70] | NA [4.93 to 4.93] — Could not be estimated due to insufficient number of events. | NA [2.23 to 2.23] — Could not be estimated due to insufficient number of events.

18. Secondary Outcome: Relapse Free Survival (RFS)
Description: RFS is defined as time from conforming JCAR017 infusion to the first progressive disease (PD), relapsed disease or death from any cause, whichever occurs first. Disease progression is defined as increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. Relapsed disease is defined as Reappearance of blasts in the blood or bone marrow (> 5%) or > 1% with previous/supportive molecular findings or in any extramedullary site after a CR. CR is defined as absence of circulating blasts, extramedullary disease, lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement, Trilineage hematopoiesis (TLH) and < 5%, Absolute neutrophil count (ANC) > 1000 per microliter, Platelets > 100,000 per microliter and no recurrence for 4 weeks.
Time Frame: Up to approximately 15 months
Population: Efficacy Analysis Set included all participants who fulfilled all study eligibility criteria, received conforming JCAR017 infusion, who did not demonstrate morphological remission at screening and who are not MRD negative upon restaging prior to initiation of lymphodepleting (LD) chemotherapy. Only responders are included in he analysis. Censored participants were also analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 4 | 1
months | 7.77 [0.46 to 14.62] | 6.98 [1.15 to 8.97] | NA [3.12 to 3.12] — Could not be estimated due to insufficient number of events.

19. Secondary Outcome: Event Free Survival (EFS)
Description: EFS is defined as time from conforming JCAR017 infusion to progressive disease (PD), relapsed disease, start of a new anticancer therapy including HSCT or death from any cause, whichever occurs first. Disease progression is defined as increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. Relapsed disease is defined as Reappearance of blasts in the blood or bone marrow (> 5%) or > 1% with previous/supportive molecular findings or in any extramedullary site after a CR. CR is defined as absence of circulating blasts, extramedullary disease, lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement, Trilineage hematopoiesis (TLH) and < 5%, Absolute neutrophil count (ANC) > 1000 per microliter, Platelets > 100,000 per microliter and no recurrence for 4 weeks. Only responders are included in he analysis. Censored participants were also analyzed.
Time Frame: From conforming JCAR017 infusion to PD, relapsed disease, start of a new anticancer therapy including Hematopoietic Stem Cell Transplant (HSCT) or death from any cause, whichever occurs first (Up to approximately 15 months)
Population: Efficacy Analysis Set included all participants who fulfilled all study eligibility criteria, received conforming JCAR017 infusion, who did not demonstrate morphological remission at screening and who are not MRD negative upon restaging prior to initiation of lymphodepleting (LD) chemotherapy. Disease assessments reported after a PD or relapsed disease were not considered for the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 4 | 1
months | 3.24 [0.46 to 14.62] | 5.42 [1.15 to 8.97] | 3.12 [3.12 to 3.12]

20. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval from the date of first confirming JCAR017 infusion to the date of death due to any reason.
Time Frame: From the date of first confirming JCAR017 infusion to the date of death due to any reason (Up to approximately 24 months)
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 4 | 1
months | 7.13 [0.76 to NA] — Could not be estimated due to insufficient number of events. | 7.08 [4.99 to NA] — Could not be estimated due to insufficient number of events. | 8.90 [NA to NA] — Could not be estimated due to insufficient number of events.

21. Secondary Outcome: Minimal Residual Response (MRD) Negative Response Rate
Description: Minimal Residual Disease (MRD) Negative Response Rate is defined as the percentage of participants achieving either a CR or CRi with a MRD negative bone marrow on Day 28, confirmed on Day 56. CR is defined as absence of circulating blasts, extramedullary disease, lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement, Trilineage hematopoiesis (TLH) and < 5%, Absolute neutrophil count (ANC) > 1000 per microliter, Platelets > 100,000 per microliter and no recurrence for 4 weeks. CRi is defined as meeting all criteria for CR except platelets < 100,000/μL or ANC is < 1000/μL. Disease progression is defined as increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. Disease assessments recorded on or after start of a new anticancer therapy, including HSCT, will not be considered, nor will disease assessments reported after a PD or relapse has been observed.
Time Frame: Up to Day 56
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 6 | 4 | 1
percentage of participants | 16.7 [0.4 to 64.1] | 25.0 [0.6 to 80.6] | 100.0 [2.5 to 100.0]

22. Secondary Outcome: Number of Participants Who Achieved a Response After JCAR017 Infusion and Then Proceeded to Hematopoietic Stem Cell Transplant
Description: Number of participants who undergo HSCT after receiving a JCAR017 infusion and achieving a response are presented. The time of proceeding to HSCT is defined as the time of commencing the conditioning regimen as required for HSCT. CR is defined as absence of circulating blasts, extramedullary disease, lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement, Trilineage hematopoiesis (TLH) and < 5%, Absolute neutrophil count (ANC) > 1000 per microliter, Platelets > 100,000 per microliter and no recurrence for 4 weeks. CRi is defined as meeting all criteria for CR except platelets < 100,000/μL or ANC is < 1000/μL. Disease progression is defined as increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease.
Time Frame: Up to approximately 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg
Number analyzed (Participants) | 7 | 6 | 1
Participants | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from JCAR017 infusion until their study completion (up to approximately 1928 days). Serious and non-serious adverse events were collected from first JCAR017 infusion (Day 1) to 90 days post JCAR017 infusion.
Description: All-cause mortality was collected for all participants that underwent leukapheresis. Serious and non-serious adverse events were collected for all participants who received conforming JCAR017 infusion. Data for Serious and Non-Serious Adverse Events was not collected for participant in the Not Assigned arm.
Arm/Group | 0.05 x 10^6 CAR+ T Cells/kg | 0.15 x 10^6 CAR+ T Cells/kg | 0.50 x 106 CAR+T Cells/kg | Not Assigned
All-Cause Mortality (participants affected / at risk) | 6/9 | 4/8 | 1/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 5/7 | 3/6 | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.05 x 10^6 CAR+ T Cells/kg (N=7) | 0.15 x 10^6 CAR+ T Cells/kg (N=6) | 0.50 x 106 CAR+T Cells/kg (N=1) | Not Assigned (N=0)
Cytokine release syndrome (Immune system disorders) | 0 | 3 | 0 | NA
Pneumonia (Infections and infestations) | 1 | 0 | 0 | NA
Sepsis (Infections and infestations) | 1 | 0 | 0 | NA
Viraemia (Infections and infestations) | 1 | 0 | 0 | NA
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | NA
Neurotoxicity (Nervous system disorders) | 1 | 1 | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.05 x 10^6 CAR+ T Cells/kg (N=7) | 0.15 x 10^6 CAR+ T Cells/kg (N=6) | 0.50 x 106 CAR+T Cells/kg (N=1) | Not Assigned (N=0)
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 1 | NA
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA
Leukopenia (Blood and lymphatic system disorders) | 4 | 1 | 1 | NA
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 1 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3 | 1 | NA
Bradycardia (Cardiac disorders) | 0 | 1 | 1 | NA
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | NA
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | NA
Anaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | NA
Anal fissure (Gastrointestinal disorders) | 1 | 1 | 0 | NA
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | NA
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | NA
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | NA
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | NA
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1 | 0 | NA
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | NA
Pyrexia (General disorders) | 1 | 0 | 0 | NA
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | NA
Cytokine release syndrome (Immune system disorders) | 4 | 1 | 1 | NA
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1 | 0 | NA
Hypogammaglobulinaemia (Immune system disorders) | 1 | 1 | 1 | NA
Bacteraemia (Infections and infestations) | 1 | 1 | 0 | NA
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | NA
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | NA
Paronychia (Infections and infestations) | 1 | 0 | 0 | NA
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | NA
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | NA
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | NA
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA
Alanine aminotransferase increased (Investigations) | 4 | 0 | 1 | NA
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 0 | NA
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0 | NA
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | NA
Blood creatinine increased (Investigations) | 1 | 0 | 0 | NA
Blood fibrinogen decreased (Investigations) | 1 | 0 | 0 | NA
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | NA
Blood uric acid increased (Investigations) | 1 | 0 | 0 | NA
Gamma-glutamyltransferase increased (Investigations) | 4 | 0 | 0 | NA
Interleukin level increased (Investigations) | 0 | 1 | 0 | NA
International normalised ratio increased (Investigations) | 1 | 0 | 0 | NA
Oxygen saturation decreased (Investigations) | 0 | 2 | 0 | NA
Serum ferritin increased (Investigations) | 0 | 1 | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | NA
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | NA
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA
Dizziness (Nervous system disorders) | 0 | 1 | 0 | NA
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | NA
Neurotoxicity (Nervous system disorders) | 0 | 1 | 1 | NA
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | NA
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | NA
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA
Cyanosis (Vascular disorders) | 0 | 1 | 0 | NA
Hypertension (Vascular disorders) | 1 | 0 | 1 | NA

LIMITATIONS AND CAVEATS:
The study was terminated and hence participants were not enrolled in Phase 2 cohorts (r/r B-ALL; MRD+ B-ALL; r/r B-NHL).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT03743246/Prot_SAP_000.pdf